CLINICAL TRIAL: NCT05963672
Title: Assessment of Sleep Quality of Hospitalized Patients Treated With EEG-guided Protection Procedures: Application in Intensive Care Unit. (SleepScan)
Brief Title: Assessment of Sleep Quality of Hospitalized Patients Treated With EEG-guided Protection Procedures: Application in Intensive Care Unit
Acronym: SleepScan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SleepScan
Record Dates: First submitted 2023-06-19; First posted 2023-07-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sleep Quality; Critically Ill Patient; Intensive Care Unit
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Sham Comparator)
  Interventions: Other: Control condition
- EEG-guided sleep protection (Experimental)
  Interventions: Device: EEG-guided sleep protection

INTERVENTIONS:
Device: EEG-guided sleep protection — The tablet will display a specific picture "prioritize sleep" or "prioritize care" depending on the patient status determined by the algorithm. When the picture "favor/prioritize sleep" is displayed, all caregivers and visiting family are asked to follow the sleep protection rules: refrain to enter the room for not urgent reasons, switch off television, reduced light in the room/corridor, reduce noise in front of the door, close curtain (if any), and delay non urgent care…etc; if caregivers have to enter the room, headlight and/or additional light will be favored. All these rules will be established collegially by nurses and doctors. Obviously, urgent care and reactions to alarms are maintained.
  When the picture "favor/prioritize care" is displayed, all caregivers and visiting family are invited to perform non urgent care, cleaning, restocking perfusion needles, comfort care, visiting.
  Arms: EEG-guided sleep protection
Other: Control condition — the recording device will be placed on the patient to record sleep but the tablet will be masked and placed face down on the bench in the room, invisible from the door.
  Arms: Usual Care

SUMMARY:
Sleep of critically ill patients is highly disturbed with a high sleep fragmentation; patients spend most of their sleep in very short sleep episodes, lasting less than 10 minutes. Causes of theses sleep alterations are complex including environmental noise (alarms, beepers, conversations…), continuous light, nurse care and repetitive measures of vital parameters.

Numerous studies have reported a relationship between severe sleep alterations and a prolonged weaning period and mortality. Improving sleep quality in critically ill patients is a major challenge to promote ICU patient's recovery.

A very promising treatment is the application of a nocturnal " quiet-time " during which non urgent care, comfort care, systematic measures of vital parameters are delayed and clustered in order to limit room entries. However, " quiet time " procedures have failed to improve sleep quality to date.

A miniaturized medical device recording one EEG channel and embedding an automated sleep scoring algorithm running in real-time was devised. This device (positioned on forehead, and continuously recording noise and light levels) indicates if the patient is awake or asleep using a tablet positioned at doorstep of the room, so that nurses know if patient is sleeping, without entering the room.

Hypothesis proposes that applying sleep protection procedures (clustering cares, limiting room entries, reducing lights and noise, delaying non urgent care…) when patients are sleeping (= EEG-guided strategies) will increase patients sleep quality.

This study will assess the effect of such device on sleep quality in ICU patients. This is a "before / after" design. The first group ("control group"), will be recorded but the sleep scoring will not be displayed by the tablet and patient will be expose to standard care. Then, procedure will be established collegially with nurses, nurses assistants and doctors. Then, the second group ("treated group") will be recorded with the device displaying the status of the patient (asleep/awake) and all caregivers will be asked to follow the established rules ("EEG-guided sleep protection rules")

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted in medical ICU of University Hospital of Poitiers

  * Un-sedated patients displaying a RASS scale between -2 and +1
  * Intubated or spontaneously breathing patients
  * Patient or family have signed the inform consent

Exclusion Criteria:

* Patients with a central nervous system disease altering sleep scoring
* Patients who received drugs (<24h) modifying significantly EEG and sleep scoring
* Patients with cutaneous erosion of the scalp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Day 1 to Day 4
  Proportion of continuous sleep

SECONDARY OUTCOMES:
Sleep fragmentation | Day 1 to Day 4
  Number of awakenings and micro-awakenings per hour of sleep
Environmental noise and environmental light | Day 1 to Day 4
  Number of peak noise end time spent above 20 lux
Sleep interruptions by caregivers | Day 1 to Day 4
  Number of room entries while patient is asleep
Sleep quality | Day 2 to Day 4
  Proportion of continuous sleep
Workload assessed by nurses | Day 1 to Day 4
  Score at specific scale assessing workload. From 1- no workload to 10- significant additional workload.
Patient Agitation | Day 1 to day 4
  Number of patients with diminishing (-1 point) Richmond Agitation-Sedation Scale (RASS) score. 10 Agitation-Sedation scale items From +4 (combative) to -5 (non-recoverable)
Performance of the algorithm | Day 1 to Day 4
  Number of sleep episodes lasting more than 10 min correctly identified by algorithm (versus vision scoring)
Patient reported sleep quality | Day 1 to day 4
  Score et richards-Campbell sleep questionnaire. It consist of 6 questions, each question scored from 0 to 100. Higher score mean the better sleep
Anxiety level | Day 1 to day 4
  Score at Spielberger Y-A scale.It consist of 12 questions, each rated on a scale with 4 response options. Lower score means a minimal anxiety level.
Respiratory status | At Unit care discharge, an average of 14 days
  Weaning duration (number of days), ventilator free days and respiratory status at discharge
Presence of delirium | Day 1 to Day 4
  Number of days with positive Confusion Assessment Method(CAM)-ICU scale. It is made up of 4 criteria. The test is POSITIVE (confusion present) if 1 and 2 + 3 or 4 are met.
Unit Care length of stay | At Unit care discharge, an average of 14 days
  Number of days in ICU
Safety of the procedure | One day after Unit Care discharge, an average of 15 days
  Numbers of Serious adverse events and Material defect events
Sleep continuity | Day 1 to Day 4
  Part of sleep time past in more than 10 minutes episodes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France